CLINICAL TRIAL: NCT00257816
Title: A Pilot Study of Weekly IV Topotecan and Cisplatin With Concurrent Pelvic Radiation in the Treatment of Stages IB2 - IVA Cervical Carcinoma
Brief Title: Weekly IV Topotecan and Cisplatin With Radiation in Cervical Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Chao Family Comprehensive Cancer Center, Cancer Center, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 03-33; 2003-3394 (Other: University of California Irvine)
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Topotecan; Cisplatin
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Topotecan; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topotecan (Experimental): Adding weekly topotecan to cisplatin in patients with primary, locally advanced carcinoma of the cervix receiving pelvic irradiation.
  Interventions: Drug: Topotecan; Drug: Cisplatin

INTERVENTIONS:
Drug: Topotecan — (First stage of accrual, 6 patients)-2 mg/m2 IV on days 1, 8, 15, 22, 29 and once during parametrial boost (6 cycles)
  If none or 1 of the 6 patients in the first Stage of accrual finish the prescribed therapy in over 8 weeks, then the second Stage of accrual (an additional 6 patients) will increase the Topotecan dose to 3 mg/m2 on days 1, 8, 15, 22, 29 and once during parametrical boost (6 cycles). If 2 or 3 of the patients in the first stage of accrual finish the prescribed therapy in over 8 weeks, the dose of the Topotecan will remain the same in the second Phase of accrual. If 4 or more of the patients in the first stage of accrual finish the prescribed therapy in over 8 weeks, there will be no second phase of accrual.
  Other Names: Hycamtin
Drug: Cisplatin — 40 mg/m2 IV (Maximum total dose of 70 mg) on days 1, 8, 15, 22, 29 and once during parametrial boost (6 cycles)
  Other Names: Platinol; AQ; NSC #119875

SUMMARY:
There will be approximately 14,000 new patients with invasive cervical cancer diagnosed in the United States in 2003 with about 4,000 deaths from this disease. This accounts for approximately 17% of all deaths due to gynecologic cancers. Radiation has been the primary treatment modality for locoregionally advanced cervical cancer. Recent trials of concomitant systemic cisplatin chemotherapy and radiation have shown high response rates (RR) with improvements in durable remissions and overall survival. Though the incidence and mortality in the U.S. dropped steadily from years 1940 to 2000, there has recently been a plateau, arresting the decline. With the routine addition of systemic Cisplatin (CDDP) chemotherapy to local regional radiation, mortality from advanced cervical cancer in the United States is expected to further decrease. However, further advances in this disease are needed.

DETAILED DESCRIPTION:
All eligible patients with invasive squamous cell, adenocarcinoma, or adenosquamous carcinoma of the cervix, Stages I-B2, II-B, III-B, and IV-A, will experience clinical staging as permitted by FIGO staging criteria.

Primary Objective:

Feasibility and toxicity of administering weekly Topotecan among patients with carcinoma of the cervix receiving concurrent pelvic radiation and Cisplatin.

Secondary Objective(s):

To assess the efficacy of administering weekly Topotecan to patients with carcinoma of the cervix receiving concurrent pelvic radiation and Cisplatin on:

* progression-free survival,
* overall survival, and
* local control

Statistic This is a feasibility study. A two phase accrual will be utilized. If none or 1 of the 6 patients in the first Stage of accrual finish the prescribed therapy in over 8 weeks, then the second Stage of accrual (an additional 6 patients) will increase the Topotecan dose to 3 mg//m2 on days 1, 8, 15, 22, 29 and once during parametrial boost (6 cycles). If 2 or 3 of the patients in the first stage of accrual finish the prescribed therapy in over 8 weeks, the dose of the Topotecan will remain the same in the second Phase of accrual. If 4 or more of the patients in the first stage of accrual finish the prescribed therapy in over 8 weeks, there will be no second phase of accrual.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary, previously untreated, histologically confirmed invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix, Stage I-2, II-B, III-B, IV-A.
2. Patients with negative, non-suspicious para-aortic nodes determined by lymphangiogram, CT, MRI or lymphadenectomy.
3. Patients with adequate bone marrow function: ANC greater than or equal to 1,500/mcl, platelets greater than or equal to 100,000/mcl, and Hemoglobin > 10 mg/dl.
4. Patients with adequate renal function: Creatinine equal to or less than 1.5 mg%.
5. Patients with adequate hepatic function: Bilirubin less than or equal to 1.5 x normal and SGOT and Alkaline phosphatase less than or equal to 3 x normal.
6. Patients who have signed an approved informed consent.
7. Patients with GOG Performance Status of 0, 1, 2, or 3.
8. Patients of childbearing potential must have a negative serum pregnancy test and use an effective form of contraception.
9. Patients who are suitable for treatment with radical intent using concurrent cisplatin and pelvic radiation.

Exclusion Criteria:

1. Patients who cannot be or have not been adequately clinically staged.
2. Patients with lower one-third vaginal involvement.
3. Patients with septicemia or severe infection.
4. Patients with circumstances that will not permit completion of the study or required follow-up.
5. Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of the other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy.
6. Patients with carcinoma of the cervical stump.
7. Patients who are lactating or pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12-17 (Actual); Study Completion 2007-12-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants in which topotecan improves response rate (RR) when added to cisplatin in treating metastatic and recurrent cervical cancer | 5 years
  Topotecan improves response rate (RR), progression-free survival (PFS) and overall survival (OS) when added to cisplatin in treating metastatic and recurrent cervical cancer. The objective of this study was to assess the feasibility of adding weekly topotecan to cisplatin in patients with primary, locally advanced carcinoma of the cervix receiving pelvic irradiation.

SECONDARY OUTCOMES:
Number of Participants in which topotecan improves progression-free survival (PFS) when added to cisplatin in treating metastatic and recurrent cervical cancer. | 5 years
  Patients will be followed clinically for evidence of tumor progression. Progression-free survival will be defined as the time from Day 1 to the date of progression or death due to any cause. Overall survival time will be measured from Day 1 until death.
Number of Participants in which topotecan improves overall survival (OS) when added to cisplatin in treating metastatic and recurrent cervical cancer. | 5 years
  OS will be assessed by clinical laboratory tests, physical examinations, vital sign measurements and the incidence and severity of adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Monk, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

REFERENCES:
- [Result] Gatcliffe TA, Tewari KS, Shah A, Brewster WR, Burger RA, Kuo JV, Monk BJ. A feasibility study of topotecan with standard-dose cisplatin and concurrent primary radiation therapy in locally advanced cervical cancer. Gynecol Oncol. 2009 Jan;112(1):85-9. doi: 10.1016/j.ygyno.2008.09.029. Epub 2008 Nov 1. PMID 18977518